CLINICAL TRIAL: NCT06197464
Title: FLOAT Through Anxiety: Examining the Efficacy and Safety of the Virtual Reality Application "Float" as a Tool to Distract From Negative Emotions and Thoughts in People With High Levels of Anxiety and Stress
Brief Title: FLOAT Through Anxiety: Virtual Reality Application's Efficacy as a Tool to Distract From Negative Emotions and Thoughts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Responsible Party: Principal Investigator, Yael Enav, Dr. Yael Enav, University of Haifa
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: YAEL
Record Dates: First submitted 2023-06-13; First posted 2024-01-09 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Control; Experimental

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Active Comparator): psychoeducation on emotional regulation and distraction strategy + Application
  Interventions: Behavioral: psychoeducation on emotional regulation and distraction strategy + Application
- experimental (Experimental): psychoeducation on emotional regulation and distraction strategy + Application with the FLOAT app
  Interventions: Behavioral: psychoeducation on emotional regulation and distraction strategy; Device: Using the FLOAT app on a virtual reality device

INTERVENTIONS:
Behavioral: psychoeducation on emotional regulation and distraction strategy — The experimenter gives the subject psychoeducation about emotional regulation and distraction strategy with the help of a conversation and a presentation.
  Arms: experimental
Device: Using the FLOAT app on a virtual reality device — The subject should wear the VR device, and use the FLOAT application.
  Arms: experimental
Behavioral: psychoeducation on emotional regulation and distraction strategy + Application — psychoeducation on emotional regulation and distraction strategy + Application
  Arms: control

SUMMARY:
The goal of this clinical trial is to examine the effectiveness and safety of the VR FLOAT application as a tool to reduce negative thoughts and feelings and anxiety symptoms in students with high levels of stress and anxiety. The main questions it aims to answer are:

1. Will subjects with high levels of anxiety who will use the FLOAT application experience a more significant relief in feelings of anxiety compared to subjects in the control group?
2. Will subjects who are used to using technology find greater comfort in using VR compared to subjects who are not used to it?
3. What is the degree of satisfaction with the use of VR and are there any reports of side effects?Participants will [describe the main tasks participants will be asked to do, treatments they'll be given and use bullets Researchers will compare control group to see The comparison between using FLOAT as a regulation strategy after psychoeducation on emotional regulation and cognitive-behavioral use of a regulation strategy after the same psychoeducation

ELIGIBILITY:
Inclusion Criteria:

* 'moderate' or 'severe' levels of stress and/or anxiety according to the DASS-21 questionnaire
* student

Exclusion Criteria:

* under the age of 18
* diagnoses of schizophrenia or bipolar disorder, including past or present psychotic conditions
* suicidality
* pregnant women
* do not speak or read Hebrew fluently
* a diagnosis of epilepsy.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2023-03-12 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2024-01-20 (Actual)

PRIMARY OUTCOMES:
situational anxiety before session | a week
  The State-Trait Anxiety Inventory (STAI) questionnaire. range 20 to 100, with a higher score representing higher levels of anxiety
situational anxiety after session | a week
  The State-Trait Anxiety Inventory (STAI) questionnaire. range 20 to 100, with a higher score representing higher levels of anxiety
satisfaction with life | baseline
  Satisfaction with Life Scale (SWLS). 5 to 35. A high score represents higher life satisfaction and a lower score represents a lower life satisfaction
satisfaction with life | week 3, after intervention
  Satisfaction with Life Scale (SWLS). 5 to 35. A high score represents higher life satisfaction and a lower score represents a lower life satisfaction
Ease of using the technology | week 3, after intervention
  System Usability Scale (SUS). scale from 0 to 100. A score higher than 70 indicates good usability, while a score lower than 50 indicates low usability.

SECONDARY OUTCOMES:
The FLOAT user experience | week 3, after intervention
  A semi-structured interview, will be analyzed qualitatively

CONTACTS AND LOCATIONS:
Overall Officials: YAEL ENAV, professor, Principal Investigator — University of Haifa
Locations (1):
- University of Haifa, Haifa, Israel